CLINICAL TRIAL: NCT04143776
Title: Renal- and Pulmonary Function in Relation to Abdominal Hypertension After Abdominal Reconstruction: The REPARE-study
Brief Title: Renal- and Pulmonary Function in Relation to Abdominal Hypertension After Abdominal Reconstruction
Acronym: REPARE
Status: Withdrawn | Type: Observational
Why Stopped: Currently on standby until new primary investigator is found
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Sinor Soltanizadeh, Medical Doctor, Ph.D.-student, Bispebjerg Hospital
Other Study IDs: 1
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Hernia, Ventral; Hernia Incisional; Acute Kidney Injury; Restrictive Lung Disease; Intraabdominal Hypertension
Keywords: hernia; abdominal reconstruction; intraabdominal pressure; acute kidney injury; restrictive lung disease
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia; Acute Kidney Injury; Intra-Abdominal Hypertension; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Abdominal reconstruction — No restrictions are set on surgical procedures or anaesthetic management.

SUMMARY:
An incisional hernia is technically challenging to operate and is the most frequent long-term complication after open surgery, resulting in impaired quality of life and reduced physical ability. Large hernias contain large amounts of abdominal volume, which similarly are missing from the abdominal cavity. Due to adaptations of the abdominal wall muscles and decreased space in the abdominal cavity, abdominal wall reconstruction lead to increased tension and thereby increased intraabdominal pressure.

Reduced renal and lung function after surgery is one of the leading causes of prolonged hospitalization, increased costs and mortality. Elevated intraabdominal pressure is a known risk factor for kidney injury, but relationships between hernia surgery, increased intraabdominal pressure, renal and lung function are still unclear.

Therefore, in patients undergoing surgery for incisional hernia, we will investigate the extent and consequences of elevated intraabdominal pressure, as well as its relation to renal injury and reduced lung function. We will also investigate the relationship between hernia dimensions and the development of increased intraabdominal pressure, as well as identifying patients at particular risk of developing elevated intraabdominal pressure.

From April 2020 to October 2021, we will include 100 patients at Bispebjerg Hospital, Denmark, diagnosed with medium to giant incisional hernia, who will undergo scheduled surgery. Patients are followed from before to 30 days after surgery. They will be examined with CT scans before and after surgery. Blood tests, pulmonary function tests and measurement intraabdominal pressure will be performed before and until 3 days after surgery. Thirty days after surgery, lung function tests and blood tests are repeated at a final examination at the out-patient clinic. During follow-up, differences in hospital stay, complications, reoperations, and mortality will be investigated.

Participation in the project is not associated with any side effects and risks. The study is expected great scientific gain, as the results can help identify particularly vulnerable patients in need of extended observation and treatment. The results obtained by the project are sought to be published in relevant scientific journals and conferences. The project is expected to extend over a 3-year period, which will include commissioning, data collection, analytical processing, dissemination of results and conduction of PhD thesis.

DETAILED DESCRIPTION:
Introduction Incisional hernia is the most common long-term complication following abdominal surgery with an estimated incidence of 10.3% within 24 months. Large incisional hernias are associated with patient discomfort, reduced quality of life and are surgically challenging with increased risks of postoperative complications. Constant contraction of the lateral abdominal wall muscles may cause displacement of a greater proportion of the abdominal contents through the hernia defect, thereby reducing volume in the abdominal cavity (loss of domain).

Abdominal wall reconstruction in patients with loss of domain may lead to increased abdominal pressure with pressures persistently being measured above 12 mm Hg. Abdominal hypertension results in direct compression on intraabdominal vessels, which can result in oedema, reduced cardiac output and hypoxia due to hypoperfusion and reduced venous return. If intraabdominal pressures exceeds 20 mm Hg abdominal compartment syndrome occurs, leading to multiorgan failure.

Intraabdominal hypertension is additionally a known risk factor in development of acute kidney injury (AKI). A pooled incidence of AKI is estimated to 13.4% after major abdominal surgery. Development of AKI is independently recognized to be associated to increased mortality, length of stay and costs in hospitalized patients. Patients with AKI are at increased risk of developing acute coronary syndrome, heart failure and infection. Additionally, patients developing AKI after general surgery are estimated to have an eight-fold increased risk of 30-day mortality. Thus, treatment of AKI is vital, complex and time-consuming.

Intraabdominal pressures above 16 mm Hg lead to pulmonary parenchymal compression, resulting in alveolar atelectasis, pulmonary infection, decreased oxygen transport across the pulmonary capillary and decreased carbon dioxide excretion. Furthermore, elevated intraabdominal pressure to the diaphragmatic pleura may hamper diaphragmatic movement, resulting in restricted respiratory compliance with reduced forced vital capacity (FVC) but retained ratio of the forced expiratory volume within 1 second above FVC (FEV1/FVC). This condition is comparable with restrictive lung disorders.

It is possible to limit postoperative acute kidney injury and respiratory complications following intermittent intraabdominal hypertension using decompressive treatment and fluid therapy. Elevated intraabdominal pressure may ideally be limited with additional surgical procedures. However, there are few reports the relationship between abdominal wall reconstruction, intraabdominal hypertension, renal- and pulmonary function. In addition, predictive factors regarding patient characteristics, hernia dimensions and surgical procedures are still unclear. In the preoperative evaluation prior to abdominal wall reconstruction, it is important to know risks and consequences of elevated abdominal pressure. Furthermore, it is important to identify patients needing close monitoring, additional decompressing management or prophylactic surgical procedures in order to decrease costs, morbidity and mortality.

In three reports, this study evaluates intraabdominal pressure after abdominal reconstruction and its relationship to renal- and pulmonary function.

Materials and methods This is a prospective observational single-center cohort study scheduled to start in April 2020. In total, 100 patients diagnosed with medium to giant incisional hernia will be included at the surgical out-patient clinic after written and oral informed consent behind closed doors at Bispebjerg Hospital. Study follow-up is 30 days after surgery. Participants will stay admitted at the surgical department at least 3 days after surgery and subsequently discharged after sufficient postoperative recovery. All participants are invited at the out-patient clinic at postoperative day (POD) 30 for a final evaluation and data collection.

Upon inclusion, following patient characteristics are collected for all participants through a case report form:

* Age
* Gender
* Smoking status
* Height
* Weight
* ASA score
* Charlson comorbidity index
* Hernia age
* Chronic obstructive pulmonary disease
* Chronic kidney disease
* Planned procedure for abdominal reconstruction
* Number of previous abdominal operations
* Use of abdominal binder

All participants will undergo preoperative CT scans of abdomen and thorax with maximized inspiration as a part of the standardized hernia protocol with collection of following data:

* Calculated lung area in frontal plane
* Site of incisional hernia
* Maximal horizontal fascial defect
* Maximal vertical fascial defect
* Hernia volume
* Abdominal volume An additional postoperative CT scan of abdomen and thorax with maximized inspiration are performed at POD 30 to estimate changes in abdominal volume and lung area.

Additionally, preoperative venous blood samples are collected and analysed for:

* Leucocytes
* C-reactive protein
* Creatinine
* Urea
* Potassium
* Sodium
* Estimated glomerular filtration rate

On POD 1, 2, 3 and 30 venous blood samples are collected and monitored for above mentioned parameters.

In all participants, a standardized bladder catheter will be placed prior surgery and maintained until POD 3. Intraabdominal pressure is indirectly measured through the bladder pressure by use of the UnoMeter™ Abdo-Pressure™ IAP monitoring system (ConvaTec Denmark A/S). This is a precise, reproducible and validated method of monitoring the intraabdominal pressure. In accordance with recommendations from previous studies, a zero reference point is marked on the patient in the midaxillary line at the iliac crest. At each measurement the patient is placed in neutral position. No restrictions will be set on the surgical procedure or postoperative treatment. The use of component separation technique or botulinum toxin A injections will be noted. The intraabdominal pressure is measured prior surgery, after extubation, on POD 1, 2 and 3. Urine output and fluid balance are monitored at POD 1, 2 and 3.

Pulmonary function test is performed using Spirobank II Basic Spirometer. FVC and FEV1 is measured upon inclusion, on POD 1, 2, 3 and 30. Severity of pulmonary restriction is graded according to guidelines set by The American Thoracic Society. During general anaesthesia, changes in the inspiratory bronchial peak pressure (IBPP) will be monitored before and after primary fascial closure with Primus® anaesthesia workstation (Dräger Denmark A/S).

AKI is defined by guidelines set by the KDIGO AKI Guideline Work Group, including any of two following:

* increase in S-creatinine by ≥0.30 mg/dl (≥26.5 μmol/l) within 48 hours, or
* increase in S-creatinine to ≥1.5 times baseline, known or assumed to have occurred within 7 days
* decrease in urine output <0.5 ml/kg//hour for 6 hours.

Furthermore, AKI severity is staged according to following criteria:

1. S-creatinine 1.5 to 1.9 times baseline or ≥0.3 mg/dl (≥26.5 μmol/l) increase or urine output <0.5 ml/kg//hour for 6 hours to 12 hours.
2. S-creatinine 2.0 to 2.9 times baseline or urine output <0.5 ml/kg//hour for ≥12 hours.

3 S-creatinine 3.0 times baseline or increase to ≥4.0 mg/dl (≥353.6 μmol/l) or urine output <0.3 ml/kg//hour for ≥24 hours or anuria for ≥12 hours.

An epidural catheter will be placed preoperatively and maintained until POD 3. In case of inability to place an epidural catheter, bilateral transversus block will be applied. Anaesthesia will be induced using propofol, remifentanil and suxamethonium. Due to the short-lived action of suxamethonium, residual relaxation when surgery starts is absent. This will be verified using the Train-Of-Four standard muscle stimulation-relaxation evaluation.

At follow-up, following data is registered for each participant:

* Length of hospital stay
* Postoperative complications according to the Clavien-Dindo classification
* Need for intubation or treatment at the intensive care unit
* Occurrence of death within 30 days

Statistical considerations A pilot study of 30 patients underwent abdominal reconstruction for incisional hernia with pre- and postoperative measurement of intraabdominal pressure. In this study, abdominal hypertension of grade 1 or higher was found in 70% of the patients. A statistical power calculation shows that at least 88 patients must be included at an expected incidence of 70%, confidence interval of 95%, spread of +/- 10% at a selected type 1 error level of 5%. It is known that the incidence of lung complications after surgery for incisional hernia is 20% and that the incidence of AKI is 1,4%. Based on the above, it is expected that inclusion of 100 patients will be able to show clinically significant causal relationships between intraabdominal hypertension, AKI, and pulmonary complications. This is done by univariate Chi-Square test and multivariable logistic regression analysis, adjusted for the relevant confounders. In addition, associations between changes in creatinine and urea will be correlated to intraabdominal pressure by linear regression analysis, as will the results of lung function tests and volume determinations by CT scan to examine correlation to changes in intraabdominal pressure.

Side effects, risks and disadvantages Placement of a bladder catheter for measurement of intraabdominal pressure is a part of the standardized hernia protocol. The bladder catheter is usually removed on POD 1, but will instead be maintained until POD 3. This is considered to be associated with a small risk of catheter-associated urinary tract infection, which will be treated according to national guidelines. Measurement of intraabdominal pressure is safe and not associated with any additional risk. On POD 1-3, venous blood samples will be drawn from each participant. This is associated with little to no pain and a considerable small risk of a small haematoma. Study participants undergo one additional CT scans within the study period. The participants are thus subjected to extra ionizing radiation. The effective participant dose is approximately 2.6 mSv per scan. By this, participants are subjected to radiation at a level which is estimated to increase the life-time risk of radiation-induced cancer by less than 0.01%. This is not considered clinically relevant. There are no other side effects, risks and disadvantages associated with participation in the study.

Respect for physical and mental integrity as well privacy This is a public research study which is reported through the regional joint notification to the Danish Data Protection agency. Information about participants is protected via the law on handling of personal information and the Danish health Act. Information about previous surgery, concurrent diseases and contact information is passed from the participants' medical charts. This information will be used to identify possible study participants. After study completion, no more information is gathered from the patient's medical chart. In case of need for further information, Sinor Soltanizadeh can contact the participant after the study is finalized. This study has been reported to the Danish National Data Protection Agency.

Economy Study initiator and primary investigator Sinor Soltanizadeh does not receive any other financial support than the salary paid by departments of which he is working full-time. The study is not company sponsored. Sinor Soltanizadeh is not associated with private sources of funding with interests in the study. No financial support is expected for this study, as the study will be departmentally funded. If support is given, the Ethical Committee of the Capital Region (RegionH) will be notified and study material including patient information will be updated.

Remuneration and other services Remuneration and other services are not paid to study participants.

Information accessibility Further information about the study is available to participants by direct inquiry to Sinor Soltanizadeh by telephone or e-mail.

Publication of results Results - positive, negative or inconclusive - will be published in relevant scientific peer-review journals, as well as presented to relevant scientific conferences. In case publication in a journal is not achieved, results will be publicly available via http://www.clinicaltrials.gov/.

Research ethics outline The overall aim of this study is to estimate the incidence of AKI and pulmonary impairment, and investigate consequences thereof in patients undergoing abdominal reconstruction. Additionally, to determine prognostic factors of developing AKI and pulmonary impairment. The participants will contribute to understanding the development AKI and pulmonary impairment. It is clinically relevant to minimize the risk of AKI, and knowledge gained from present study will help to understand preventive measures in certain patients. Participants are expected to gain from this study by a more thorough monitoring of their renal function and pulmonary function and gain access to earlier necessary treatment.

Participation in this study is considered to be associated to minimal risks and side effects. The autonomy as well as the integrity of the participant is not compromised in any way by participating in the study.

In conclusion, this study is considered to be in concordance with ethical standards, as the possible gain from participation exceeds the risks associated.

Recruitment of participants Patients are recruited at the out-patient clinic of Bispebjerg Hospital at the time of first contact. In case a patient fulfils in- and exclusion criteria, they are informed about the study and given oral and written participant information. Patients will be informed of their right to have an assessor present at the time of information. The information will be given in a private room where the door is closed in order to avoid disturbance. Patients are offered one week of consideration time before deciding whether or not to participate in the study, and will be offered a new interview for after the consideration time. In case patients themselves declare they need no time to reflect, oral and written consent can be given immediately after the first information is given.

ELIGIBILITY:
Inclusion Criteria:

* Horizontal fascial defects of >8 cm defined by preoperative CT scan
* Planned elective open incisional hernia repair

Exclusion Criteria:

* Pregnancy
* Previous bladder resection or reconstruction
* Chronic catheter use
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with medium to giant incisional hernia undergoing planned open incisional hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Intraabdominal hypertension after abdominal reconstruction | Before surgery, on postoperative day 1, 2 and 3.
  The primary aim is to investigate changes in the intraabdominal pressure after abdominal reconstruction.
Pulmonary function in intraabdominal hypertension after abdominal reconstruction | Before surgery, on postoperative day 30.
  The primary aim is to investigate changes in the pulmonary areal after abdominal reconstruction through pre- and postoperative CT scans.
Surgical complications and intraabdominal hypertension after abdominal reconstruction | From surgery to postoperative day 30.
  The primary aims are to estimate length of stay in patients with and without intraabdominal hypertension.

SECONDARY OUTCOMES:
Intraabdominal hypertension after abdominal reconstruction | Before surgery, on postoperative day 1, 2 and 3.
  Secondary aims are to estimate the risk of intraabdominal hypertension in correlation with loss of domain defined by preoperative CT scans and to estimate the incidence of AKI in patients with and without intraabdominal hypertension.
Pulmonary function in intraabdominal hypertension after abdominal reconstruction | Before surgery, during surgery, on postoperative day 1, 2, 3 and 30.
  Secondary aims are to investigate immediate intraoperative changes in inspiratory peak pressures before and after primary fascial closure and estimate the incidence of postoperative restrictive pulmonary dysfunction.
Surgical complications and intraabdominal hypertension after abdominal reconstruction | From surgery to postoperative day 30. Predicting factors are assessed preoperatively.
  Secondary aims are to investigate complications, reoperations and 30-day mortality in patients with and without intraabdominal hypertension. Furthermore, to evaluate predicting factors of intraabdominal hypertension in relation to hernia dimensions, comorbidities and surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sinor Soltanizadeh, MD, Principal Investigator — Digestive Disease Center, Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Digestive Disease Center, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Will be determined later.

REFERENCES:
- [Background] Itatsu K, Yokoyama Y, Sugawara G, Kubota H, Tojima Y, Kurumiya Y, Kono H, Yamamoto H, Ando M, Nagino M. Incidence of and risk factors for incisional hernia after abdominal surgery. Br J Surg. 2014 Oct;101(11):1439-47. doi: 10.1002/bjs.9600. Epub 2014 Aug 14. PMID 25123379
- [Background] Jensen KK, Munim K, Kjaer M, Jorgensen LN. Abdominal Wall Reconstruction for Incisional Hernia Optimizes Truncal Function and Quality of Life: A Prospective Controlled Study. Ann Surg. 2017 Jun;265(6):1235-1240. doi: 10.1097/SLA.0000000000001827. PMID 27280505
- [Background] Kokotovic D, Bisgaard T, Helgstrand F. Long-term Recurrence and Complications Associated With Elective Incisional Hernia Repair. JAMA. 2016 Oct 18;316(15):1575-1582. doi: 10.1001/jama.2016.15217. PMID 27750295
- [Background] Parker SG, Halligan S, Blackburn S, Plumb AAO, Archer L, Mallett S, Windsor ACJ. What Exactly is Meant by "Loss of Domain" for Ventral Hernia? Systematic Review of Definitions. World J Surg. 2019 Feb;43(2):396-404. doi: 10.1007/s00268-018-4783-7. PMID 30187090
- [Background] Petro CC, Raigani S, Fayezizadeh M, Rowbottom JR, Klick JC, Prabhu AS, Novitsky YW, Rosen MJ. Permissible Intraabdominal Hypertension following Complex Abdominal Wall Reconstruction. Plast Reconstr Surg. 2015 Oct;136(4):868-881. doi: 10.1097/PRS.0000000000001621. PMID 26090761
- [Background] Malbrain ML, De Laet IE, De Waele JJ, Kirkpatrick AW. Intra-abdominal hypertension: definitions, monitoring, interpretation and management. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):249-70. doi: 10.1016/j.bpa.2013.06.009. PMID 24012236
- [Background] Cheatham ML. Abdominal compartment syndrome: pathophysiology and definitions. Scand J Trauma Resusc Emerg Med. 2009 Mar 2;17:10. doi: 10.1186/1757-7241-17-10. PMID 19254364
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Background] Demarchi AC, de Almeida CT, Ponce D, e Castro MC, Danaga AR, Yamaguti FA, Vital D, Gut AL, Ferreira AL, Freschi L, Oliveira J, Teixeira UA, Christovan JC, Grejo JR, Martin LC. Intra-abdominal pressure as a predictor of acute kidney injury in postoperative abdominal surgery. Ren Fail. 2014 May;36(4):557-61. doi: 10.3109/0886022X.2013.876353. Epub 2014 Jan 23. PMID 24456177
- [Background] O'Connor ME, Kirwan CJ, Pearse RM, Prowle JR. Incidence and associations of acute kidney injury after major abdominal surgery. Intensive Care Med. 2016 Apr;42(4):521-530. doi: 10.1007/s00134-015-4157-7. Epub 2015 Nov 24. PMID 26602784
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Biteker M, Dayan A, Tekkesin AI, Can MM, Tayci I, Ilhan E, Sahin G. Incidence, risk factors, and outcomes of perioperative acute kidney injury in noncardiac and nonvascular surgery. Am J Surg. 2014 Jan;207(1):53-9. doi: 10.1016/j.amjsurg.2013.04.006. Epub 2013 Sep 17. PMID 24050540
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] da Silva Almeida JR, Machado FS, Schettino GP, Park M, Azevedo LC. Cardiopulmonary effects of matching positive end-expiratory pressure to abdominal pressure in concomitant abdominal hypertension and acute lung injury. J Trauma. 2010 Aug;69(2):375-83. doi: 10.1097/TA.0b013e3181e12b3a. PMID 20699747
- [Background] Soltanizadeh S, Helgstrand F, Jorgensen LN. Botulinum Toxin A as an Adjunct to Abdominal Wall Reconstruction for Incisional Hernia. Plast Reconstr Surg Glob Open. 2017 Jun 21;5(6):e1358. doi: 10.1097/GOX.0000000000001358. eCollection 2017 Jun. PMID 28740773
- [Background] Nguyen DH, Nguyen MT, Askenasy EP, Kao LS, Liang MK. Primary fascial closure with laparoscopic ventral hernia repair: systematic review. World J Surg. 2014 Dec;38(12):3097-104. doi: 10.1007/s00268-014-2722-9. PMID 25145817
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Kimball EJ, Mone MC, Wolfe TR, Baraghoshi GK, Alder SC. Reproducibility of bladder pressure measurements in critically ill patients. Intensive Care Med. 2007 Jul;33(7):1195-1198. doi: 10.1007/s00134-007-0641-z. Epub 2007 Apr 28. PMID 17468849
- [Background] Cheatham ML, De Waele JJ, De Laet I, De Keulenaer B, Widder S, Kirkpatrick AW, Cresswell AB, Malbrain M, Bodnar Z, Mejia-Mantilla JH, Reis R, Parr M, Schulze R, Puig S; World Society of the Abdominal Compartment Syndrome (WSACS) Clinical Trials Working Group. The impact of body position on intra-abdominal pressure measurement: a multicenter analysis. Crit Care Med. 2009 Jul;37(7):2187-90. doi: 10.1097/CCM.0b013e3181a021fa. PMID 19487946
- [Background] Dempsey TM, Scanlon PD. Pulmonary Function Tests for the Generalist: A Brief Review. Mayo Clin Proc. 2018 Jun;93(6):763-771. doi: 10.1016/j.mayocp.2018.04.009. PMID 29866281
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Mazzocchi M, Dessy LA, Sorvillo V, Di Ronza S, Scuderi N. A study of intraabdominal pressure modification in "component separation" technique for repair of incisional hernia. Ann Ital Chir. 2010 Nov-Dec;81(6):433-7. PMID 21456479
- [Background] Blatnik JA, Krpata DM, Pesa NL, Will P, Harth KC, Novitsky YW, Rowbottom JR, Rosen MJ. Predicting severe postoperative respiratory complications following abdominal wall reconstruction. Plast Reconstr Surg. 2012 Oct;130(4):836-841. doi: 10.1097/PRS.0b013e318262f160. PMID 22691844
- [Background] Chung CU, Nelson JA, Fischer JP, Wink JD, Serletti JM, Kovach SJ. Acute kidney injury after open ventral hernia repair: an analysis of the 2005-2012 ACS-NSQIP datasets. Hernia. 2016 Feb;20(1):131-8. doi: 10.1007/s10029-015-1395-0. Epub 2015 Jun 23. PMID 26099501